CLINICAL TRIAL: NCT01841970
Title: Multi-Center, Prospective Study of the Safety and Efficacy of the HET Bipolar System for Treatment of Stage I and Stage II Hemorrhoids
Brief Title: Safety and Efficacy Study of HET Bipolar System for Treatment of Stage I and Stage II Hemorrhoids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HET-12-001
Record Dates: First submitted 2013-04-22; First posted 2013-04-29 (Estimated); Results first posted 2017-01-16 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2016-11

CONDITIONS: Hemorrhoids, Internal
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HET Arm (Other): Active arm. A single procedure with HET was used to treat Grade I and Grade II hemorrhoids
  Interventions: Device: HET Bipolar System

INTERVENTIONS:
Device: HET Bipolar System — The HET Bipolar System is used to treat hemorrhoids by bipolar ligation of the superior hemorrhoidal blood supply.

SUMMARY:
Hemorrhoids are vascular cushions in the anal canal. People are normally born with hemorrhoids, and the presence of hemorrhoids does not imply disease. However, hemorrhoids typically cause symptoms when they enlarge over time. There are two types of hemorrhoids- External Hemorrhoids and Internal Hemorrhoids.

Current minimally invasive technologies for the treatment of internal hemorrhoids are associated with several drawbacks that include high rate of recurrence and a need for repetitive procedures, frequent post-procedural pain or significant discomfort, intra-operative pain and technically demanding. The purpose of this study is to determine whether the HET Bipolar System is safe and effective in the treatment of Stage I and Stage II hemorrhoids (internal hemorrhoids). The HET Bipolar System is a new alternative device for the minimally invasive treatment of Stage I and Stage II hemorrhoids that incorporate design features with the intent of resolving each of the major limitations of currently available technology.

DETAILED DESCRIPTION:
In this study, the investigators will use the HET Bipolar System for the treatment of Stage I and Stage II hemorrhoids, where significant tissue prolapse is not present. The hemorrhoids are treated by bipolar ligation of the superior hemorrhoidal blood supply.

Each prospective subject will be screened for inclusion and exclusion criteria at least one week prior to treatment. All patients undergoing treatment will review and sign the study Informed Consent prior to their procedure.

One to three internal hemorrhoids will be treated in one therapeutic session. The number will be based on the investigator's judgment of which quadrants are symptomatic. Evaluations will be recorded for all treated subjects immediately following treatment. Subjects will be followed at 1, 3, and 6 months post procedure unless complications are reported between scheduled follow-up dates. At each post treatment follow-up, a report will be made of pain/discomfort, bleeding, medication use, itching, presence of adverse events or complications and need for supplemental treatment. Face-to-face follow-up evaluations will include anoscopic evaluation and assessment of hemorrhoid and other relevant symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Subject over 21 years of age
* General good health
* Subject undergoing elective treatment for Stage I or Stage II internal hemorrhoids
* Chronic bleeding from Stage I or Stage II internal hemorrhoids (at least weekly occurrence
* Failure of prior medical management

Exclusion Criteria:

* Under 21 years of age.
* Gastrointestinal bleeding from source other than their internal hemorrhoids
* Active proctitis
* Inflammatory bowel disease
* HIV positive or immunocompromised
* Rectal wall prolapse
* Stage III and Stage IV hemorrhoids
* Medical conditions requiring anticoagulants and/or subject to receive anticoagulants within 7 days of initial examination
* Pregnancy
* Rectal malignancy
* Hepatitis C
* Liver cirrhosis
* End stage renal disease
* Receiving chemotherapy
* Advanced malignancy
* Documented bleeding diathesis
* Treatment with an investigational drug or medical device in the past 30 days

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-04; Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- HET Arm: All subjects enrolled into the study were treated with the HET Bipolar System
Period: Overall Study
Arm/Group | HET Arm
Started | 20
Completed | 9
Not Completed | 11
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 2
Not completed — Lost to Follow-up | 8

BASELINE CHARACTERISTICS:
Arm/Group | HET Arm
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (18.1)
Gender [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 20
Hemorrhoid grade [Number; unit: participants] — Hemorrhoids as graded on a scale of I-IV, with I being least symptomatic. Grade I: Bleeding hemorrhoids which do not prolapse outside the anal canal • Grade II: Hemorrhoids which prolapse, usually with defecation, but retract spontaneously
  participants
    Grade I | 7
    Grade II | 13
Pain (Y/N) [Number; unit: participants]
  Pain Yes | 13
  Pain No | 7
Bleeding (Y/N) [Number; unit: participants]
  Bleeding Yes | 20
  Bleeding No | 0
Previous Treatment Received (Y/N) [Number; unit: participants]
  Previous Treatment Yes | 20
  Previous Treatment No | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Resolution of Symptoms
Description: The primary endpoint analysis was the resolution of symptoms, including resolution of bleeding and prolapse, if present prior to treatment
Time Frame: Post treatment at Month1, Month 3, Month 6
Population: 18 participants included. 2 participants were lost to follow up.
Measure: Number; unit: participants
Arm/Group | HET Arm
Number analyzed (Participants) | 18
participants | 18

2. Secondary Outcome: Incidence of Recurrence of Pre-procedure Symptoms
Description: Recurrence of pre-procedure symptoms after initial improvement
Time Frame: Post treatment at Month 1, Month 3, and Month 6
Measure: Number; unit: participants
Arm/Group | Month 1 | Month 3 | Month 6
Number analyzed (Participants) | 18 | 11 | 9
participants
  Recurrence Yes | 0 | 3 | 4
  Recurrence No | 18 | 8 | 5

3. Secondary Outcome: Recurrence of Symptoms That Had Resolved With Treatment
Description: Number of patients with recurrence of symptoms defined as external thrombosed hemorrhoids, infection, mucous discharge, new fissure, stenosis and delayed healing.
Time Frame: Post treatment at Month 1, Month 3, Month 6
Population: At Month 1, 3 and 6 the number of participants include patients followed through that time period. The remaining patients were lost to follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Month 1 | Month 3 | Month 6
Number analyzed (Participants) | 18 | 11 | 9
Participants
  External Thrombosed Hemorrhoids - NO | 18 | 11 | 9
  External Thrombosed Hemorrhoids - YES | 0 | 0 | 0
  Signs of Infection YES | 0 | 0 | 0
  Signs of Infection NO | 18 | 11 | 9
  Mucous Discharge YES | 0 | 0 | 0
  Mucous Discharge NO | 18 | 11 | 9
  New Fissure YES | 2 | 0 | 0
  New Fissure NO | 16 | 11 | 9
  Delayed Healing YES | 0 | 0 | 0
  Delayed Healing NO | 18 | 11 | 9
  Stenosis YES | 0 | 0 | 0
  Stenosis NO | 18 | 11 | 9
  Other Conditions YES | 2 | 2 | 1
  Other Conditions No | 15 | 9 | 8

4. Secondary Outcome: Pain Recorded Yes or No on Visual Analog Scale (VAS)
Description: Patient reported pain on 10 point scale where 0 =No Pain and > 0 = Pain with 10 being the worst.
Time Frame: Post treatment at Month 1, Month 3, Month 6
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Month 1 | Month 3 | Month 6
Number analyzed (Participants) | 18 | 11 | 9
participants
  Pain YES | 4 | 1 | 1
  Pain NO | 14 | 10 | 8

5. Secondary Outcome: Mean Pain Score Based on the Visual Analog Pain Scale
Description: Mean pain score based on the Visual Analog pain scale. Patient reported pain on 10 point scale where 0 =No Pain and > 0 = Pain with 10 being the worst.
Time Frame: Post treatment at Month 1, Month 3, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Month 1 | Month 3 | Month 6
Number analyzed (Participants) | 18 | 11 | 9
units on a scale | 0.7 (1.57) | 0.4 (1.21) | 0.1 (0.33)

ADVERSE EVENTS:
Arm/Group | HET Arm
Serious Adverse Events (participants affected / at risk) | 2/20
Other Adverse Events (participants affected / at risk) | 5/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HET Arm (N=20)
internal engorged hemorrhoids (Gastrointestinal disorders) | 1 (1) — The event was assessed as not related to the device, and was considered to be a recurrence of the study disease.
Bleeding (Gastrointestinal disorders) | 1 (1)
pain (Gastrointestinal disorders) | 1 (1)
urgency (Gastrointestinal disorders) | 1 (1)
skin tags (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HET Arm (N=20)
Bleeding/Refractory Bleeding (Gastrointestinal disorders) | 5
Gas/Gas Pain (Gastrointestinal disorders) | 2
Intermittent Burning (Gastrointestinal disorders) | 1
Internal Engorged Hemorrhoids (Gastrointestinal disorders) | 1
New Fissure (Gastrointestinal disorders) | 2
Pain (Gastrointestinal disorders) | 3
Pruritis (Gastrointestinal disorders) | 1
Recurrence (Gastrointestinal disorders) | 4
Skin Tags (Gastrointestinal disorders) | 1
Thrombosed Hemorrhoids (Gastrointestinal disorders) | 1
Urgency (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No